CLINICAL TRIAL: NCT00051298
Title: Olanzapine Versus Placebo in the Treatment of Adolescents With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4066; F1D-MC-HGIN
Record Dates: First submitted 2003-01-07; First posted 2003-01-09 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine
Drug: Placebo

SUMMARY:
This study is to determine the efficacy (how well the drug works), safety, and any side effects of olanzapine compared to placebo in the treatment of schizophrenia in adolescents. Both the potential benefits and side effects of olanzapine will be evaluated throughout this trial.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female patients, 13 to 17 years of age
* Patients must have a diagnosis of schizophrenia per DSM-IV-TR.
* Female patients of child-bearing potential must test negative for pregnancy at the time of enrollment.
* Both the patient and the patient's parent/authorized legal representative must understand the nature of the study and must sign a document granting consent.
* Patients must be capable of swallowing study medication whole (without crushing, dissolving, etc.)

Exclusion Criteria:

* Female patients who are either pregnant or nursing.
* Patients with acute or unstable medical conditions.
* Patients who have been judged clinically to be at serious suicidal risks.
* Patients who have previously not responded to an adequate dose and/or duration of olanzapine treatment.
* Patients who currently have delusional disorder, psychotic disorder NOS, schizophreniform, schizoaffective disorder, bipolar disorder, attention deficit/hyperactivity disorder or major depressive disorder.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2002-11; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of a flexible dose of olanzapine compared to placebo in the treatment of adolescents (ages 13 - 17) with schizophrenia using the BPRS-C

SECONDARY OUTCOMES:
Assess secondary efficacy measures to capture additional evidence of efficacy utilizing the CGI-I, CGI-S, PANSS and OAS
Assess the efficacy of olanzapine compared with placebo in improving clinical symptomatology in terms of rate of response
Assess the safety of olanzapine compared with placebo for up to 6 weeks of double-blind treatment and for up to an additional 26 weeks of open-label olanzapine treatment.
Assess the health-related quality of life and cognition associated with olanzapine compared with placebo for up to 6 weeks of double-blind treatment and for up to an additional 26 weeks of open-label olanzapine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, Cerritos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Hershey, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Madison, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Bellaire, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Kirkland, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hrs, EST), or speak with your personal physician., Moscow, Russia

REFERENCES:
- [Derived] Kryzhanovskaya LA, Robertson-Plouch CK, Xu W, Carlson JL, Merida KM, Dittmann RW. The safety of olanzapine in adolescents with schizophrenia or bipolar I disorder: a pooled analysis of 4 clinical trials. J Clin Psychiatry. 2009 Feb;70(2):247-58. doi: 10.4088/jcp.08m03538. Epub 2009 Feb 10. PMID 19210948
- [Derived] Kryzhanovskaya L, Schulz SC, McDougle C, Frazier J, Dittmann R, Robertson-Plouch C, Bauer T, Xu W, Wang W, Carlson J, Tohen M. Olanzapine versus placebo in adolescents with schizophrenia: a 6-week, randomized, double-blind, placebo-controlled trial. J Am Acad Child Adolesc Psychiatry. 2009 Jan;48(1):60-70. doi: 10.1097/CHI.0b013e3181900404. PMID 19057413
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com